CLINICAL TRIAL: NCT05301933
Title: A Pilot Proof of Concept, Multisite, Open Clinical Trial of Telehealth Behavioral Parent Training on Improving Access and Outcomes for Children With ADHD
Brief Title: Telehealth BPT in DBP Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-01458
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Behavioral: Behavioral Parent Training (BPT)

INTERVENTIONS:
Behavioral: Behavioral Parent Training (BPT) — BPT is an evidence-based psychosocial intervention that is directed exclusively to parent of children with ADHD and related disorders. BPT focuses on instructing parents to use approaches to enhance the parent-child relationship (e.g., quality time, praise) and proactive discipline strategies (e.g., time out, reward systems) to reduce challenging child behavior.

SUMMARY:
Access to evidence-based psychosocial interventions, particularly Behavioral Parent Training (BPT), for youth with Attention Deficit/Hyperactivity Disorder (ADHD) is limited. An approach to increasing such access is to utilize trained paraprofessionals (Family Peer Advocates; FPAs) in the delivery of BPT, particularly through modalities, like telehealth, that further improve access and availability. This approach, FPA-delivered BPT via telehealth has yet to be studied. This study will evaluate the benefits of a FPA-delivered BPT for parents of children identified with ADHD in Developmental Behavioral Pediatric (DBPs).

DETAILED DESCRIPTION:
There are two aims of the study: Specific Aim 1: To determine the benefits of a FPA-delivered telehealth BPT model on children's ADHD symptoms, oppositional behavior, functional outcomes, parenting behavior and parental stress. Specific Aim 2: Understand the shared decision making process between the parent, physician, and FPA within the Pediatric- Family Peer Advocate (PEDS-FPA) model through qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Child must be between the ages of 4-11 years
2. Child must be diagnosed with ADHD (any subtype) within the last 6 months
3. Parent/ legal guardian must be at least 18 years old
4. Parent/ legal guardian must be legal guardian of child
5. Parent/ legal guardian must speak English or Spanish
6. Parent/ legal guardian must not have previously received manualized, multi-session behavioral parent training (BPT)
7. Child must be under public or no insurance
8. Parent/legal guardian must be able to provide consent.

Exclusion Criteria:

1. Children with ADHD who have significant mental health comorbidities that warrant more intensive psychosocial/pharmacological intervention per physician recommendations
2. Parent/ legal guardian who does not have access to reliable internet service to participate in telehealth delivered BPT
3. Parent/ legal guardian with known significant impairment that will be barrier to communication and participation (e.g., intellectual disability, schizophrenia, other significant mental illness)
4. Parent/ legal guardian who has limited, consistent contact with their child (i.e., less than 3 days/week)

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Change in IOWA Connors Rating Scale (IOWA-CRS) Score | Baseline, Week 11
  The IOWA-CRS is a widely used brief measure of attention-deficit/hyperactivity disorder and oppositional-defiant behavior in children completed by parents. IOWA-CRS consists of 10 items evaluated using a four-point Likert scale with the following anchors: not at all (0); just a little (1); pretty much (2); and very much (3). The total score range is 10-40; the higher the score, the more concerns with the child's behavior.
Change in Impairment Rating Scale (IRS) Score | Baseline, Week 11
  The IRS measures impairment across domains of functioning, as well as overall need for treatment - consists of 7 items. Parents report on a 7-point scale to signify their child's functioning along a continuum of impairment that ranges from 0 (Not a problem at all. Definitely does not need treatment or special services.) to 6 (Extreme problem. Definitely needs treatment and special services). The total score range is 0-42; the higher the score, the more extreme the challenges and higher the need for intervention.
Change in Alabama Parenting Questionnaire- Short Form (APQ-9) Score | Baseline, Week 11
  APQ-9 is a well-validated 9-item measure of parenting style. Items are rated by the parent scored based on frequency of parenting behavior from Never (1), Almost Never (2), Sometimes (3), Often (4), Always (5). APQ-SF items are based around the three main structures: positive parenting (items 1, 6-7), inconsistent discipline (items 2, 4, 9) and poor supervision (items 3, 5, 8). The score range per structure is 3-27; the higher the score, the more frequent the parenting behavior (e.g., higher scores in positive parenting structure indicates more frequent positive parenting).
Change in Parental Stress - Short Form (PSI-SF) Total Stress Score | Baseline, Week 11
  PSI-SF is a 36-item self-report measure used to assess parenting stress in three domains, Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The PSI-SF is measured along a 5-point scale with one (Strongly Disagree) to five (Strongly Agree). Higher scores indicate greater levels of parenting stress. For this study, the Total Stress score, which is the sum of the three PSI-SF domains, will be used (total score range = 36-180).
Change in Barriers to Treatment Participation Scale (BTPS) Score | Baseline, Week 11
  BTPS measures barriers to treatment participation involving stressors and obstacles that compete with treatment (e.g., conflict with significant other), treatment demands and issues (e.g., treatment was too confusing), and perceived relevance of treatment (treatment met parent's expectations). BTPS consists of 18 items and is measured along a 5-point scale with 1 (Never a problem) to 5 (Always a problem). The total score range is 18-90; the higher the score, the more barriers to treatment participant.
Change in Therapy Attitude Inventory (TAI) Score | Baseline, Week 11
  TAI is a valid index of consumer satisfaction for participants in BPT. Items are rated on a scale from one (indicating treatment dissatisfaction or lack of improvement) to five (indicating satisfaction with treatment and improvement). Parents will complete this form after the last session of the BPT program. BPT consists of 11 items that are scored on a 5-point Likert scale. The total score range is 11-55; the higher the score, the greater the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hopkins, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Steinhart Department of Applied Psychology, New York, New York
  - NYU Langone Health - NYC Health+Hospitals, Bellevue Hospital, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio